CLINICAL TRIAL: NCT03560466
Title: One Year Study to Evaluate the Long-term Safety and Tolerability of Dupilumab in Pediatric Patients With Asthma Who Participated in a Previous Dupilumab Asthma Clinical Study
Brief Title: Assessment of the Safety and Efficacy of Dupilumab in Children With Asthma (Liberty Asthma Excursion)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTS14424; U1111-1200-1757 (Registry Identifier: ICTRP); 2017-003317-25 (EudraCT Number)
Record Dates: First submitted 2018-03-22; First posted 2018-06-18 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — dupilumab; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dupilumab (Experimental): Doses of dupilumab will be administered every 2 weeks or every 4 weeks added to current controller medications for 52 weeks
  Interventions: Drug: Dupilumab (SAR231893/REGN668); Drug: Asthma controller therapies (incl. prednisone/prednisolone); Drug: Asthma reliever therapies

INTERVENTIONS:
Drug: Dupilumab (SAR231893/REGN668) — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous (sc)
Drug: Asthma controller therapies (incl. prednisone/prednisolone) — Pharmaceutical form: powder, or solution, or pill
  Route of administration: inhaled, oral or parenteral
Drug: Asthma reliever therapies — Pharmaceutical form: powder or solution
  Route of administration: inhaled

SUMMARY:
Primary Objective:

* To evaluate the long-term safety and tolerability of dupilumab in pediatric patients with asthma who participated in a previous dupilumab asthma clinical study.
* To evaluate the efficacy of dupilumab in children of 6 to <12 years of age with uncontrolled persistent asthma in the Japan sub-study.

Secondary Objectives:

* To evaluate the long-term efficacy of dupilumab in pediatric patients with asthma who participated in a previous dupilumab asthma clinical study.
* To evaluate dupilumab in pediatric patients with asthma who participated in a previous dupilumab asthma clinical study with regard to:

  * Systemic exposure.
  * Anti-drug antibodies (ADAs).
  * Biomarkers.
* To evaluate the safety and tolerability of dupilumab in pediatric patients with asthma in the Japan sub-study
* To evaluate dupilumab in pediatric patients with asthma in the Japan substudy with regard to:

  * Systemic exposure,
  * Anti-drug antibodies (ADAs),
  * Biomarkers

DETAILED DESCRIPTION:
Study duration per participant is approximatively 64 weeks including a 52 weeks treatment period and 12 weeks post treatment follow-up.

Japan substudy:

Study duration per participant is approximately 68 weeks including 3-5 weeks screening period, 52 weeks treatment period and 12 weeks post treatment follow-up period.

ELIGIBILITY:
Inclusion criteria :

* Pediatric patients with asthma who completed the treatment in a dupilumab asthma trial (EFC14153).
* Signed written informed consent/assent. Specific for Brazil: EFC14153 patients from Brazil, who prematurely discontinued Investigational Medicinal Product (IMP) to receive Yellow Fever vaccine (a live attenuated vaccine) during Yellow Fever outbreak, are allowed to be enrolled in LTS14424 after completing the required procedures in EFC14153 (completion of remaining visits and procedures until end of treatment (EOT) V28, considered as V1 for LTS14424).

Patients who are not able to complete their treatment in Study EFC14153 due to the COVID-19 pandemic will be allowed to enroll into Study LTS14424. Patients who enroll in LTS14424 after completing the EFC14153 EOS visit should have eligibility for LTS14424 reevaluated including background medication check and laboratory assessments (including complete blood count [CBC] with differential and basic chemistry) within 1 month prior to LTS14424 Visit 1.

For Japan sub-study

* Signed written inform consent/assent
* Children 6 to <12 years of age, with a physician diagnosis of persistent asthma for ≥12 months prior to screening
* Blood eosinophil count ≥150 cells/μL or fractional exhaled nitric oxide (FeNO) ≥20 parts per billion (ppb) at screening visit (Visit 0).

Exclusion criteria:

* Any chronic lung disease other than asthma (eg, cystic fibrosis, bronchopulmonary dysplasia) which may impair lung function.
* Inability to follow the procedures of the study/noncompliance (eg, due to language problems or psychological disorders).
* Patients receiving concomitant treatment or required a new concomitant treatment prohibited in the study.
* Patients or his/her parent(s)/caregiver(s)/legal guardian(s) is related to the Investigator or any Sub-Investigator, research assistant, pharmacist, study coordinator, other staff thereof directly involved in the conduct of the study.
* Patients who experienced any hypersensitivity reactions to dupilumab in a previous dupilumab study, which, in the opinion of the Investigator, could indicate that continued treatment with dupilumab may present an unreasonable risk for the patient.
* Any abnormalities or adverse events at screening (last treatment visit in the study EFC14153 will be the screening visit) that per Investigator judgment would adversely affect patient's participation in this study or would require permanent IMP discontinuation.
* For female patients who have commenced menstruating at any time during the study and are either:
* Found to have a positive urine pregnancy test, or
* Sexually active, not using an established acceptable contraceptive method.
* Planned live, attenuated vaccinations during the study.
* Patients with active autoimmune disease or patients using immunosuppressive therapy for autoimmune disease (eg, juvenile idiopathic arthritis, inflammatory bowel disease, systemic lupus erythematosus) at enrollment.

For Japan sub-study:

* Any chronic lung disease other than asthma (eg, cystic fibrosis, bronchopulmonary dysplasia) which may impair lung function.
* Inability to follow the procedures of the study/noncompliance (eg, due to language problems or psychological disorders).
* Patients receiving concomitant treatment or required a new concomitant treatment prohibited in the study at the screening and enrollment visits.
* Patients who previously have been treated with dupilumab
* Diagnosed with active parasitic infection (helminthes); suspected or high risk of parasitic infection, unless clinical and (if necessary) laboratory assessments have ruled out active infection before randomization
* Known or suspected history of immunosuppression, including history of invasive opportunistic infections (eg, histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, aspergillosis), despite infection resolution; or unusually frequent, recurrent, or prolonged infections, per Investigator's judgment.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 378 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (81):
- United States (12):
  - Arizona Allergy and Immunology Research- Site Number : 8400002, Gilbert, Arizona
  - Asthma and Airway Disease Research Center Site Number : 8400012, Tucson, Arizona
  - Peninsula Research Associates Site Number : 8400001, Rolling Hills Estates, California
  - Division of Pulmonary Medicine and Allergy Medicine- Site Number : 8400006, St Louis, Missouri
  - Somnos Clinical Research Site Number : 8400022, Lincoln, Nebraska
  - Northwell Health- Site Number : 8400023, Great Neck, New York
  - Columbia University Medical Center- Site Number : 8400013, New York, New York
  - Rochester Regional Health- Site Number : 8400007, Rochester, New York
  - Immunocarolina LLC Site Number : 8400004, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center Site Number : 8400008, Cincinnati, Ohio
  - OK Clinical Research, LLC- Site Number : 8400024, Edmond, Oklahoma
  - Allergy & Asthma Research Center- Site Number : 8400003, San Antonio, Texas
- Argentina (5):
  - Investigational Site Number : 0320002, CABA, Buenos Aires
  - Investigational Site Number : 0320001, CABA, Buenos Aires
  - Investigational Site Number : 0320004, Vicente Lopez, Buenos Aires F.D.
  - Investigational Site Number : 0320003, Buenos Aires
  - Investigational Site Number : 0320006, Mendoza
- Investigational Site Number : 0360005, North Adelaide, South Australia, Australia
- Brazil (5):
  - Irmandade da Santa Casa de Misericordia de Porto Alegre- Site Number : 0760001, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas da PUCRS- Site Number : 0760007, Porto Alegre, Rio Grande do Sul
  - Unidade Ambulatorial de Pesquisa Clinica I - NGP - UNIFESP- Site Number : 0760002, São Paulo, São Paulo
  - Instituto da Criança of Hospital das Clínicas de São Paulo- Site Number : 0760004, São Paulo, São Paulo
  - Clinica de Alergia Martti Antila Site Number : 0760006, Sorocaba, São Paulo
- Investigational Site Number : 1240003, Québec, Canada
- Chile (5):
  - Investigational Site Number : 1520001, Valdivia, Los Ríos Region
  - Investigational Site Number : 1520005, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520009, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520007, Viña del Mar, Región de Valparaíso
  - Investigational Site Number : 1520002, Viña del Mar, Región de Valparaíso
- Colombia (2):
  - Investigational Site Number : 1700004, Antioquia
  - Investigational Site Number : 1700002, Cali
- Hungary (7):
  - Investigational Site Number : 3480006, Budapest
  - Investigational Site Number : 3480002, Gyula
  - Investigational Site Number : 3480012, Mezőkövesd
  - Investigational Site Number : 3480001, Székesfehérvár
  - Investigational Site Number : 3480008, Szigetvár
  - Investigational Site Number : 3480003, Töröbálint
  - Investigational Site Number : 3480007, Zalaegerszeg
- Italy (3):
  - Investigational Site Number : 3800003, Florence
  - Investigational Site Number : 3800004, Padua
  - Investigational Site Number : 3800005, Roma
- Japan (11):
  - Investigational Site Number : 3920013, Chiba, Chiba
  - Investigational Site Number : 3920016, Chuo-ku, Chiba
  - Investigational Site Number : 3920005, Yotsukaido-shi, Chiba
  - Investigational Site Number : 3920015, Fukuoka, Fukuoka
  - Investigational Site Number : 3920011, Fukuoka, Fukuoka
  - Investigational Site Number : 3920008, Shibukawa, Gunma
  - Investigational Site Number : 3920014, Onomichi-shi, Hiroshima
  - Investigational Site Number : 3920003, Sapporo, Hokkaido
  - Investigational Site Number : 3920012, Tsu, Mie-ken
  - Investigational Site Number : 3920010, Ureshino-shi, Saga-ken
  - Investigational Site Number : 3920009, Habikino-Shi
- Lithuania (4):
  - Investigational Site Number : 4400005, Šiauliai
  - Investigational Site Number : 4400003, Utena
  - Investigational Site Number : 4400001, Vilnius
  - Investigational Site Number : 4400004, Vilnius
- Mexico (5):
  - Investigational Site Number : 4840006, Chihuahua City
  - Investigational Site Number : 4840004, Chihuahua City
  - Investigational Site Number : 4840003, Durango, Durango
  - Investigational Site Number : 4840001, Monterrey, Nuevo León
  - Investigational Site Number : 4840002, Veracruz
- Poland (2):
  - Investigational Site Number : 6160002, Poznan, Greater Poland Voivodeship
  - Investigational Site Number : 6160001, Lodz, Lódzkie
- Russia (5):
  - Investigational Site Number : 6430004, Perm
  - Investigational Site Number : 6430002, Saint Petersburg
  - Investigational Site Number : 6430001, Saint Petersburg
  - Investigational Site Number : 6430003, Saint Petersburg
  - Investigational Site Number : 6430005, Saint Petersburg
- Investigational Site Number : 7100001, Cape Town, South Africa
- Investigational Site Number : 7240001, Barcelona, Barcelona [Barcelona], Spain
- Turkey (Türkiye) (4):
  - Investigational Site Number : 7920005, Adana
  - Investigational Site Number : 7920001, Ankara
  - Investigational Site Number : 7920003, Istanbul
  - Investigational Site Number : 7920004, Istanbul
- Ukraine (7):
  - Investigational Site Number : 8040007, Chernivtsi
  - Investigational Site Number : 8040004, Dnipro
  - Investigational Site Number : 8040005, Kharkiv
  - Investigational Site Number : 8040008, Kryvyi Rig
  - Investigational Site Number : 8040001, Kyiv
  - Investigational Site Number : 8040002, Zaporizhzhya
  - Investigational Site Number : 8040003, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Bacharier LB, Maspero JF, Katelaris CH, Fiocchi AG, Gagnon R, de Mir I, Guilbert TW, Jackson DJ, Staudinger HW, Laws E, Mannent LP, Akinlade B, Maloney J, Tawo K, Khokhar FA, Li N, Hardin M, Abdulai RM, Lederer DJ, Robinson LB; Liberty Asthma EXCURSION Investigators. Assessment of long-term safety and efficacy of dupilumab in children with asthma (LIBERTY ASTHMA EXCURSION): an open-label extension study. Lancet Respir Med. 2024 Jan;12(1):45-54. doi: 10.1016/S2213-2600(23)00303-X. Epub 2023 Nov 10. PMID 37956679

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The main study was conducted at 70 centers in 17 countries, and the sub-study was conducted at 11 centers in Japan. 365 participants who rolled over from parent study EFC14153 (NCT02948959) were enrolled in the main study and 13 participants (not included in parent study EFC14153) were enrolled in Japan sub-study.
Pre-assignment Details: All participants received dupilumab dose based on body weight in the main study and Japan sub-study. As pre-specified in the protocol and statistical analysis plan (SAP), the results are presented by study and treatment group, regardless of the dose regimen.
Groups:
- Main Study: Placebo-Dupilumab: Participants who received placebo matched to dupilumab in the parent study EFC14153 received dupilumab for 52 weeks in the main study as follows:
  * 100 milligrams (mg) once every 2 weeks (q2w) as a subcutaneous (SC) injection or 300 mg once every 4 weeks (q4w) as an SC injection for participants with body weight ≤30 kilograms (kg).
  * 200 mg q2w as an SC injection for participants with body weight >30 kg. Participants also received a stable-dose background therapy of medium-dose inhaled corticosteroids (ICS) with a second controller medication (i.e., long-acting beta-2 agonists [LABA], long-acting muscarinic antagonists [LAMA], leukotriene receptor antagonists [LTRA] or methylxanthines) or high-dose ICS alone or high-dose ICS with second controller medication. Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication as instructed by Investigator.
- Main Study: Dupilumab-Dupilumab: Participants who received dupilumab in the parent study EFC14153 received dupilumab for 52 weeks in the main study as follows:
  * 100 mg q2w as an SC injection or 300 mg q4w as an SC injection for participants with body weight ≤30 kg.
  * 200 mg q2w as an SC injection for participants with body weight >30 kg. Participants also received a stable-dose background therapy of medium-dose ICS with a second controller medication (i.e., LABA, LAMA, LTRA or methylxanthines) or high-dose ICS alone or high-dose ICS with second controller medication. Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication as instructed by Investigator.
- Japan Sub-study: Dupilumab: Participants received dupilumab for 52 weeks in the Japan sub-study as follows:
  * 100 mg q2w as an SC injection or 300 mg q4w as an SC injection for participants with body weight ≥15 kg and ≤30 kg.
  * 200 mg q2w as an SC injection for participants with body weight >30 kg. Participants also received a stable-dose background therapy of medium-dose ICS with a second controller medication (i.e., LABA, LAMA, LTRA or methylxanthines) or high-dose ICS alone or high-dose ICS with second controller medication. Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication as instructed by Investigator.
Period: Overall Study
Arm/Group | Main Study: Placebo-Dupilumab | Main Study: Dupilumab-Dupilumab | Japan Sub-study: Dupilumab
Started | 125 | 240 | 13
Completed | 118 | 228 | 12
Not Completed | 7 | 12 | 1
Not completed — Adverse Event | 1 | 2 | 0
Not completed — Poor Compliance to Protocol | 0 | 2 | 0
Not completed — Other | 6 | 8 | 1

BASELINE CHARACTERISTICS:
Population: Main study: safety population included all participants exposed to at least 1 dose or part of a dose of the study treatment during current study regardless of the amount of treatment administered. Sub-study: enrolled population included all participants who signed the informed consent/assent and had a treatment kit number allocated and recorded in the interactive voice response system/interactive web response system database, regardless of whether the treatment kit was received or not.
Groups:
- Main Study: Placebo-Dupilumab: Participants who received placebo matched to dupilumab in the parent study EFC14153 received dupilumab for 52 weeks in the main study as follows:
  * 100 mg q2w as an SC injection or 300 mg q4w as an SC injection for participants with body weight ≤30 kg.
  * 200 mg q2w as an SC injection for participants with body weight >30 kg. Participants also received a stable-dose background therapy of medium-dose ICS with a second controller medication (i.e., LABA, LAMA, LTRA or methylxanthines) or high-dose ICS alone or high-dose ICS with second controller medication. Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication as instructed by Investigator.
- Total: Total of all reporting groups
Arm/Group | Main Study: Placebo-Dupilumab | Main Study: Dupilumab-Dupilumab | Japan Sub-study: Dupilumab | Total
Number analyzed (Participants) | 125 | 240 | 13 | 378
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.9 (1.6) | 9.9 (1.7) | 9.69 (1.11) | 9.89 (1.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 85 | 4 | 135
  Male | 79 | 155 | 9 | 243
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/White | 111 | 215 | 0 | 326
  Black/of African Descent | 6 | 9 | 0 | 15
  Asian | 0 | 1 | 13 | 14
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Other | 8 | 14 | 0 | 22

OUTCOME MEASURES:

1. Primary Outcome: Main Study: Number of Participants With Any Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. TEAEs were AEs that developed or worsened or became serious during the TEAE period.
Time Frame: From first dose of study treatment (Day 1) up to 112 days post last dose of study treatment, approximately 64 weeks
Population: Safety population included all participants exposed to at least 1 dose or part of a dose of the study treatment during current study regardless of the amount of treatment administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Placebo-Dupilumab | Main Study: Dupilumab-Dupilumab
Number analyzed (Participants) | 125 | 240
Participants | 85 | 147

2. Primary Outcome: Japan Sub-study: Change From Baseline to Week 12 in Pre-Bronchodilator Percent Predicted Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 was the volume of air (in liters) exhaled from the lungs in the first second of a forced expiration as measured by spirometer. Spirometry was performed after a wash out period of bronchodilators according to their action duration. Baseline was defined as the last available measurement prior to the first study treatment dose if the participant was treated, or the last available value up to enrollment if the participant was not exposed to study treatment in the current study.
Time Frame: Baseline (Day 1) to Week 12
Population: Intent-to-treat (ITT) population included all participants in the enrolled population in the current study.
Measure: Mean (Standard Deviation); unit: percent predicted FEV1
Arm/Group | Japan Sub-study: Dupilumab
Number analyzed (Participants) | 13
percent predicted FEV1 | 7.08 (6.78) [lower limit 6.78]

3. Secondary Outcome: Japan Sub-study: Number of Participants With Any Treatment-Emergent Adverse Events
Description: An AE was any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. TEAEs were AEs that developed or worsened or became serious during the TEAE period.
Time Frame: From first dose of study treatment (Day 1) up to 112 days post last dose of study treatment, approximately 64 weeks
Population: Safety population included all enrolled participants who took at least 1 dose of study treatment in the current study, regardless of the amount of treatment administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Japan Sub-study: Dupilumab
Number analyzed (Participants) | 13
Participants | 13

4. Secondary Outcome: Annualized Rate of Severe Asthma Exacerbation Events During the 52-Week Treatment Period
Description: A severe exacerbation event during study was defined as a deterioration of asthma requiring use of systemic corticosteroid (SCS) for ≥3 days or hospitalization/emergency room visit because of asthma, requiring SCS. Annualized severe exacerbation event rate was defined as total number of events that occurred during 52-week treatment period divided by total number of participant-years followed in 52-week treatment period.
Time Frame: Up to Week 52
Population: Main study: safety population included all participants exposed to at least 1 dose or part of a dose of study treatment during current study regardless of amount of treatment administered. Sub-study: ITT population included all participants in enrolled population in the current study.
Measure: Number; unit: exacerbations per participant-years
Arm/Group | Main Study: Placebo-Dupilumab | Main Study: Dupilumab-Dupilumab | Japan Sub-study: Dupilumab
Number analyzed (Participants) | 125 | 240 | 13
exacerbations per participant-years | 0.114 | 0.120 | 0.462

5. Secondary Outcome: Change From Baseline in Pre-Bronchodilator Percent Predicted Forced Expiratory Volume in 1 Second Over Time
Description: FEV1 was volume of air (in liters) exhaled from the lungs in first second of a forced expiration as measured by spirometer. Spirometry was performed after a wash out period of bronchodilators according to their action duration. Baseline (main study): original baseline of parent study EFC14153. Baseline (sub-study): last available measurement prior to first study treatment dose if participant was treated, or last available value up to enrollment if participant was not exposed to study treatment in current study.
Time Frame: Baseline (Day 1) and Weeks 2, 4 (Japan sub-study), 8, 12, 24, 52 and 64
Population: Main study: safety population included all participants exposed to at least 1 dose or part of a dose of study treatment during current study regardless of amount of treatment administered. Sub-study: ITT population included all participants in enrolled population in current study. Only participants with data collected at the specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: percent predicted FEV1
Arm/Group | Main Study: Placebo-Dupilumab | Main Study: Dupilumab-Dupilumab | Japan Sub-study: Dupilumab
Number analyzed (Participants) | 122 | 231 | 13
percent predicted FEV1
  Week 2: number analyzed (Participants) | 122 | 231 | 12
  Week 2 | 8.06 (15.71) | 11.03 (18.74) | 7.50 (9.29)
  Week 4: number analyzed (Participants) | 0 | 0 | 13
  Week 4 |  |  | 7.00 (7.12)
  Week 8: number analyzed (Participants) | 120 | 222 | 13
  Week 8 | 7.93 (14.88) | 12.47 (18.60) | 6.31 (8.97)
  Week 12: number analyzed (Participants) | 118 | 226 | 13
  Week 12 | 8.31 (14.70) | 10.95 (17.33) | 7.08 (6.78)
  Week 24: number analyzed (Participants) | 118 | 219 | 13
  Week 24 | 8.37 (15.48) | 11.23 (18.24) | 4.08 (8.75)
  Week 52: number analyzed (Participants) | 116 | 212 | 11
  Week 52 | 8.81 (16.18) | 12.19 (17.88) | 6.73 (8.09)
  Week 64: number analyzed (Participants) | 112 | 212 | 12
  Week 64 | 7.98 (17.14) | 10.67 (17.19) | 1.17 (8.03)

6. Secondary Outcome: Change From Baseline in Absolute Forced Expiratory Volume in 1 Second Over Time
Description: as for outcome 5
Time Frame: Baseline (Day 1) and Weeks 2, 4 (Japan sub-study), 8, 12, 24, 52 and 64
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Main Study: Placebo-Dupilumab | Main Study: Dupilumab-Dupilumab | Japan Sub-study: Dupilumab
Number analyzed (Participants) | 122 | 231 | 13
liter
  Week 2: number analyzed (Participants) | 122 | 231 | 12
  Week 2 | 0.36 (0.32) | 0.42 (0.38) | 0.13 (0.15)
  Week 4: number analyzed (Participants) | 0 | 0 | 13
  Week 4 |  |  | 0.13 (0.13)
  Week 8: number analyzed (Participants) | 120 | 222 | 13
  Week 8 | 0.38 (0.32) | 0.47 (0.39) | 0.12 (0.15)
  Week 12: number analyzed (Participants) | 118 | 226 | 13
  Week 12 | 0.41 (0.31) | 0.45 (0.36) | 0.17 (0.13)
  Week 24: number analyzed (Participants) | 118 | 219 | 13
  Week 24 | 0.46 (0.35) | 0.51 (0.39) | 0.15 (0.15)
  Week 52: number analyzed (Participants) | 116 | 212 | 11
  Week 52 | 0.62 (0.41) | 0.66 (0.41) | 0.34 (0.21)
  Week 64: number analyzed (Participants) | 112 | 212 | 12
  Week 64 | 0.66 (0.45) | 0.70 (0.44) | 0.25 (0.14)

7. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) Over Time
Description: FVC was defined as volume of air (in liters) that could be forcibly blown out after full inspiration in upright position as measured by spirometer. Spirometry was performed after wash out period of bronchodilators according to their action duration. Baseline (main study):original baseline of parent study EFC14153. Baseline (sub-study): last available measurement prior to first study treatment dose if participant was treated or last available value up to enrollment if participant was not exposed to study treatment in current study.
Time Frame: Baseline (Day 1) and Weeks 2, 4 (Japan sub-study), 8, 12, 24, 52 and 64
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Main Study: Placebo-Dupilumab | Main Study: Dupilumab-Dupilumab | Japan Sub-study: Dupilumab
Number analyzed (Participants) | 122 | 231 | 13
liter
  Week 2: number analyzed (Participants) | 122 | 231 | 12
  Week 2 | 0.35 (0.29) | 0.38 (0.38) | 0.11 (0.15)
  Week 4: number analyzed (Participants) | 0 | 0 | 13
  Week 4 |  |  | 0.09 (0.12)
  Week 8: number analyzed (Participants) | 120 | 222 | 13
  Week 8 | 0.37 (0.30) | 0.45 (0.42) | 0.11 (0.14)
  Week 12: number analyzed (Participants) | 118 | 226 | 13
  Week 12 | 0.40 (0.30) | 0.43 (0.39) | 0.12 (0.11)
  Week 24: number analyzed (Participants) | 118 | 219 | 13
  Week 24 | 0.47 (0.36) | 0.50 (0.40) | 0.17 (0.15)
  Week 52: number analyzed (Participants) | 116 | 212 | 11
  Week 52 | 0.68 (0.42) | 0.70 (0.45) | 0.36 (0.22)
  Week 64: number analyzed (Participants) | 112 | 212 | 12
  Week 64 | 0.74 (0.49) | 0.75 (0.48) | 0.41 (0.24)

8. Secondary Outcome: Change From Baseline in Forced Expiratory Flow [FEF] 25% to 75% Over Time
Description: FEF was defined as amount of air which can be forcibly exhaled from lungs in first second of forced exhalation. FEF 25-75% was the mean FEF between 25% and 75% of FVC. FVC was defined as volume of air that could be forcibly blown out after full inspiration in upright position. Spirometry was performed after wash out period of bronchodilators. Baseline (main study): original baseline of parent study EFC14153. Baseline (sub-study): last available measurement prior to first study treatment dose if participant was treated or last available value up to enrollment if participant was not exposed to study treatment in current study.
Time Frame: Baseline (Day 1) and Weeks 2, 4 (Japan sub-study), 8, 12, 24, 52 and 64
Population: Main study: safety population included all participants exposed to at least 1 dose or part of dose of study treatment during current regardless of amount of treatment administered. Sub-study: ITT population included all participants in enrolled population in current study. Only participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: liter per second
Arm/Group | Main Study: Placebo-Dupilumab | Main Study: Dupilumab-Dupilumab | Japan Sub-study: Dupilumab
Number analyzed (Participants) | 122 | 231 | 13
liter per second
  Week 2: number analyzed (Participants) | 122 | 231 | 12
  Week 2 | 0.49 (0.63) | 0.58 (0.66) | 0.21 (0.26)
  Week 4: number analyzed (Participants) | 0 | 0 | 13
  Week 4 |  |  | 0.25 (0.23)
  Week 8: number analyzed (Participants) | 120 | 222 | 13
  Week 8 | 0.48 (0.60) | 0.62 (0.63) | 0.15 (0.30)
  Week 12: number analyzed (Participants) | 118 | 226 | 13
  Week 12 | 0.54 (0.60) | 0.59 (0.61) | 0.29 (0.31)
  Week 24: number analyzed (Participants) | 118 | 219 | 13
  Week 24 | 0.58 (0.68) | 0.66 (0.65) | 0.15 (0.37)
  Week 52: number analyzed (Participants) | 116 | 212 | 11
  Week 52 | 0.73 (0.75) | 0.77 (0.67) | 0.40 (0.46)
  Week 64: number analyzed (Participants) | 112 | 212 | 12
  Week 64 | 0.77 (0.78) | 0.79 (0.70) | 0.11 (0.34)

9. Secondary Outcome: Main Study: Change From Baseline in Percent Predicted Forced Vital Capacity Over Time
Description: FVC was defined as volume of air (in liters) that could be forcibly blown out after full inspiration in upright position as measured by spirometer. Spirometry was performed after wash out period of bronchodilators according to their action duration. Baseline was defined as the original baseline of parent study EFC14153.
Time Frame: Baseline (Day 1) and Weeks 2, 8, 12, 24, 52 and 64
Population: Safety population included all participants exposed to at least 1 dose or part of a dose of study treatment during current study regardless of amount of treatment administered. Only participants with data collected at the specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: percent predicted FVC
Arm/Group | Main Study: Placebo-Dupilumab | Main Study: Dupilumab-Dupilumab
Number analyzed (Participants) | 122 | 231
percent predicted FVC
  Week 2 | 2.98 (12.91) | 5.02 (16.33)
  Week 8: number analyzed (Participants) | 120 | 222
  Week 8 | 2.88 (12.17) | 6.64 (17.42)
  Week 12: number analyzed (Participants) | 118 | 226
  Week 12 | 3.23 (12.49) | 5.03 (16.45)
  Week 24: number analyzed (Participants) | 118 | 219
  Week 24 | 3.19 (13.35) | 5.28 (16.20)
  Week 52: number analyzed (Participants) | 116 | 212
  Week 52 | 3.74 (13.10) | 6.43 (16.40)
  Week 64: number analyzed (Participants) | 112 | 212
  Week 64 | 3.13 (15.14) | 4.83 (16.09)

10. Secondary Outcome: Japan Sub-study: Change From Baseline in Asthma Control Questionnaire-Interviewer Administered, 7-Question Version (ACQ-7-IA) Over Time
Description: ACQ-7-IA had 7 questions with first 5 items of ACQ-7 addressing most common asthma symptoms: frequency in past week awoken by asthma during night, severity of asthma symptoms in morning, limitation of daily activities due to asthma, shortness of breath due to asthma, wheeze; 2 questions on short-acting bronchodilator use and predicted bronchodilator use of FEV1. Participants/parents/guardians recalled child's previous week asthma and responded to questions on 7-point scale: 0=no impairment, 6=maximum impairment. Global ACQ-7-IA score was the mean of 7 questions, ranging from 0 (totally controlled) to 6 (severely uncontrolled). Higher scores indicated lower asthma control. Baseline: last available measurement prior to first study treatment dose if participant was treated or last available value up to enrollment if participant was not exposed to study treatment in current study.
Time Frame: Baseline (Day 1) and Weeks 2, 4, 8, 12, 24, 36, 52 and 64
Population: ITT population included all participants in enrolled population in current study. Only participants with data collected at specified timepoints are reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Japan Sub-study: Dupilumab
Number analyzed (Participants) | 13
score on a scale
  Week 2 | -0.65 (0.64)
  Week 4 | -0.68 (0.75)
  Week 8 | -0.84 (0.59)
  Week 12 | -1.03 (0.66)
  Week 24 | -0.96 (0.61)
  Week 36 | -1.01 (0.47)
  Week 52 | -1.21 (0.37)
  Week 64: number analyzed (Participants) | 12
  Week 64 | -0.99 (0.52)

11. Secondary Outcome: Japan Sub-study: Change From Baseline in Asthma Control Questionnaire-Interviewer Administered, 5-Question Version (ACQ-5-IA) Over Time
Description: The ACQ-5-IA had 5 questions addressing most common asthma symptoms: frequency in past week awoken by asthma during night, severity of asthma symptoms in morning, limitation of daily activities due to asthma, shortness of breath due to asthma and wheeze. Participants/parents/guardians recalled the child's previous week asthma and responded to symptom and bronchodilator use questions on a 7-point scale: 0=no impairment, 6=maximum impairment. Global ACQ-5-IA score was the mean of 5 questions, ranging from 0 (totally controlled) to 6 (severely uncontrolled). Higher score indicated lower asthma control. Baseline: last available measurement prior to first study treatment dose if participant was treated, or last available value up to enrollment if participant was not exposed to study treatment in current study.
Time Frame: Baseline (Day 1) and Weeks 2, 4, 8, 12, 24, 36, 52 and 64
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Japan Sub-study: Dupilumab
Number analyzed (Participants) | 13
score on a scale
  Week 2 | -0.68 (0.87)
  Week 4 | -0.75 (1.06)
  Week 8 | -0.92 (0.82)
  Week 12 | -1.20 (0.84)
  Week 24 | -1.15 (0.68)
  Week 36 | -1.25 (0.54)
  Week 52 | -1.49 (0.54)
  Week 64: number analyzed (Participants) | 12
  Week 64 | -1.28 (0.59)

12. Secondary Outcome: Serum Concentrations of Dupilumab
Description: Blood samples were collected at the specified timepoints for determination of functional dupilumab concentration in serum.
Time Frame: Weeks 12, 24, 52 and 64
Population: Pharmacokinetic population:participants in safety population with atleast 1 nonmissing;evaluable predose serum concentration post 1st dose of dupilumab in current study.Only participants with data collected at specified timepoints are reported.As prespecified in SAP,serum concentration is presented by dose regimen.Main study:dose regimen was adjusted per participant's weight during study,hence some participants may be counted in more than 1 dose regimen across different weeks based on weight.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Groups:
- Main Study: Dupilumab 100 mg q2w: All participants from the main study who received dupilumab 100 mg q2w were included in this arm.
- Main Study: Dupilumab 200 mg q2w: All participants from the main study who received dupilumab 200 mg q2w were included in this arm.
- Main Study: Dupilumab 300 mg q4w: All participants from the main study who received dupilumab 300 mg q4w were included in this arm.
- Japan Sub-study: Dupilumab 100 mg q2w: All participants from the Japan sub-study who received dupilumab 100 mg q2w were included in this arm.
- Japan Sub-study: Dupilumab 200 mg q2w: All participants from the Japan sub-study who received dupilumab 200 mg q2w were included in this arm.
- Japan Sub-study: Dupilumab 300 mg q4w: All participants from the Japan sub-study who received dupilumab 300 mg q4w were included in this arm.
Arm/Group | Main Study: Dupilumab 100 mg q2w | Main Study: Dupilumab 200 mg q2w | Main Study: Dupilumab 300 mg q4w | Japan Sub-study: Dupilumab 100 mg q2w | Japan Sub-study: Dupilumab 200 mg q2w | Japan Sub-study: Dupilumab 300 mg q4w
Number analyzed (Participants) | 52 | 299 | 16 | 3 | 7 | 3
nanogram per milliliter
  Week 12: number analyzed (Participants) | 52 | 296 | 6 | 3 | 7 | 3
  Week 12 | 60740.38 (23885.77) | 80450.15 (39865.24) | 79600.00 (25509.84) | 38600.00 (20850.18) | 79128.57 (24513.31) | 53066.67 (18569.96)
  Week 24: number analyzed (Participants) | 38 | 293 | 12 | 3 | 6 | 3
  Week 24 | 64201.03 (22890.02) | 81849.66 (42824.93) | 80675.00 (26921.27) | 41300.00 (22138.65) | 98316.67 (18066.81) | 55166.67 (14558.96)
  Week 52: number analyzed (Participants) | 27 | 299 | 16 | 3 | 7 | 3
  Week 52 | 52808.85 (21526.05) | 71910.74 (42290.54) | 81289.94 (31957.07) | 41000.00 (23157.94) | 91128.57 (28739.33) | 59300.00 (18107.46)
  Week 64: number analyzed (Participants) | 28 | 298 | 16 | 3 | 6 | 3
  Week 64 | 1884.04 (9763.01) | 3391.86 (16196.36) | 184.69 (582.75) | 39.00 (0.00) | 39.00 (0.00) | 39.00 (0.00)

13. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADAs) Against Dupilumab
Description: ADA positive was defined as either treatment-boosted or treatment-emergent response in the ADA assay. Treatment-boosted response was defined as a positive response in the ADA assay post first dose in the current study that was greater than or equal to 4-fold of the baseline titer levels, when baseline results were positive. Treatment-emergent response was defined as a positive response in the ADA assay post first dose in the current study, when baseline results were negative or missing. Baseline (main study): original baseline of parent study EFC14153. Baseline (sub-study): last available measurement prior to first study treatment dose if participant was treated, or last available value up to enrollment if participant was not exposed to study treatment in current study.
Time Frame: From first dose of study treatment (Day 1) to Week 64
Population: ADA population (main and sub-study) included all the participants in the safety population with at least 1 non-missing ADA result following the first dose of dupilumab in the current study. Only participants with data collected for the specified categories are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Placebo-Dupilumab | Main Study: Dupilumab-Dupilumab | Japan Sub-study: Dupilumab
Number analyzed (Participants) | 124 | 239 | 13
Participants
  Treatment-boosted ADA Response: number analyzed (Participants) | 2 | 3 | 0
  Treatment-boosted ADA Response | 1 | 0 |
  Treatment-emergent ADA Response: number analyzed (Participants) | 122 | 236 | 13
  Treatment-emergent ADA Response | 10 | 7 | 2

14. Secondary Outcome: Main Study: Percent Change From Baseline in Blood Eosinophil Count at Week 64
Description: Blood samples were collected at specified timepoints to assess percent change from baseline in eosinophil count. Baseline was defined as the original baseline of parent study EFC14153.
Time Frame: Baseline (Day 1) to Week 64
Population: Safety population included all participants exposed to at least 1 dose or part of a dose of the study treatment during current study regardless of the amount of treatment administered. Only participants with data collected are reported.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Main Study: Placebo-Dupilumab | Main Study: Dupilumab-Dupilumab
Number analyzed (Participants) | 103 | 186
percent change | 34.528 (207.067) [lower limit 207.067] | 29.769 (323.837) [lower limit 323.837]

15. Secondary Outcome: Percent Change From Baseline in Total Immunoglobulin (Ig) E in Serum at Week 64
Description: Blood samples were collected at specified timepoints to assess percent change from baseline in total IgE in serum. Baseline (main study): the original baseline of parent study EFC14153. Baseline (sub-study): last available measurement prior to first study treatment dose if participant was treated, or last available value up to enrollment if participant was not exposed to study treatment in current study.
Time Frame: Baseline (Day 1) to Week 64
Population: Main study: safety population included all participants exposed to at least 1 dose or part of a dose of the study treatment during current study regardless of the amount of treatment administered. Sub-study: safety population included all enrolled participants who took at least 1 dose of study treatment in the current study, regardless of the amount of treatment administered. Only participants with data collected are reported.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Main Study: Placebo-Dupilumab | Main Study: Dupilumab-Dupilumab | Japan Sub-study: Dupilumab
Number analyzed (Participants) | 113 | 219 | 12
percent change | -76.9 (-85.2) [-85.2 to -63.4] | -86.8 (-91.4) [-91.4 to -77.3] | -75.0 (-81.1) [-81.1 to -70.0]

16. Secondary Outcome: Japan Sub-study: Change From Baseline in Fractional Exhaled Nitric Oxide (FeNO) at Week 64
Description: FeNO was analyzed using a NIOX instrument or similar analyzer using a flow rate of 50 milliliter per second. FeNO assessment was conducted prior to spirometry and following a fast of ≥1 hour. Baseline was defined as the last available measurement prior to first study treatment dose if participant was treated, or last available value up to enrollment if participant was not exposed to study treatment in the current study.
Time Frame: Baseline (Day 1) to Week 64
Population: Safety population included all enrolled participants who took at least 1 dose of study treatment in the current study, regardless of the amount of treatment administered. Only participants with data collected are reported.
Measure: Mean (Standard Deviation); unit: parts per billion
Arm/Group | Japan Sub-study: Dupilumab
Number analyzed (Participants) | 12
parts per billion | -8.3 (27.5) [lower limit 27.5]

ADVERSE EVENTS:
Time Frame: AEs: From first dose of study treatment (Day 1) up to 112 days post last dose of study treatment, approximately 64 weeks for main study and sub-study each. Deaths: From first dose of study treatment (Day 1) up to end of follow-up, approximately 353 weeks.
Description: Analysis was performed on safety population. As pre-specified in the protocol and SAP, the results are presented by study and treatment group, regardless of the dose regimen.
Groups:
- Main Study: Placebo-Dupilumab: Participants who received placebo matched to dupilumab in the parent study EFC14153 received dupilumab for 52 weeks in the main study as follows: - 100 mg q2w as an SC injection or 300 mg q4w as an SC injection for participants with body weight ≤30 kg. - 200 mg q2w as an SC injection for participants with body weight >30 kg. Participants also received a stable-dose background therapy of medium-dose ICS with a second controller medication (i.e., LABA, LAMA, LTRA or methylxanthines) or high-dose ICS alone or high-dose ICS with second controller medication. Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication as instructed by Investigator.
- Main Study: Dupilumab-Dupilumab: Participants who received dupilumab in the parent study EFC14153 received dupilumab for 52 weeks in the main study as follows: - 100 mg q2w as an SC injection or 300 mg q4w as an SC injection for participants with body weight ≤30 kg. - 200 mg q2w as an SC injection for participants with body weight >30 kg. Participants also received a stable-dose background therapy of medium-dose ICS with a second controller medication (i.e., LABA, LAMA, LTRA or methylxanthines) or high-dose ICS alone or high-dose ICS with second controller medication. Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication as instructed by Investigator.
- Japan Sub-study: Dupilumab: Participants received dupilumab for 52 weeks in the Japan sub-study as follows: - 100 mg q2w as an SC injection or 300 mg q4w as an SC injection for participants with body weight ≥15 kg and ≤30 kg. - 200 mg q2w as an SC injection for participants with body weight >30 kg. Participants also received a stable-dose background therapy of medium-dose ICS with a second controller medication (i.e., LABA, LAMA, LTRA or methylxanthines) or high-dose ICS alone or high-dose ICS with second controller medication. Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication as instructed by Investigator.
Arm/Group | Main Study: Placebo-Dupilumab | Main Study: Dupilumab-Dupilumab | Japan Sub-study: Dupilumab
All-Cause Mortality (participants affected / at risk) | 0/125 | 0/240 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/125 | 6/240 | 4/13
Other Adverse Events (participants affected / at risk) | 63/125 | 108/240 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study: Placebo-Dupilumab (N=125) | Main Study: Dupilumab-Dupilumab (N=240) | Japan Sub-study: Dupilumab (N=13)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Complicated Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Radius Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (5)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study: Placebo-Dupilumab (N=125) | Main Study: Dupilumab-Dupilumab (N=240) | Japan Sub-study: Dupilumab (N=13)
Eosinophilia (Blood and lymphatic system disorders) | 7 (8) | 8 (8) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dental Caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 10 (10) | 2 (3)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 5 (7) | 1 (1)
Injection Site Erythema (General disorders) | 3 (6) | 7 (11) | 1 (4)
Injection Site Induration (General disorders) | 0 (0) | 1 (2) | 1 (1)
Injection Site Reaction (General disorders) | 9 (73) | 8 (46) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 5 (5) | 6 (7)
Bronchitis (Infections and infestations) | 5 (6) | 7 (10) | 3 (4)
Covid-19 (Infections and infestations) | 1 (1) | 3 (3) | 2 (2)
Herpes Zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 7 (9) | 13 (16) | 5 (8)
Lower Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 12 (17) | 21 (25) | 5 (12)
Oral Herpes (Infections and infestations) | 1 (1) | 0 (0) | 1 (2)
Pharyngitis (Infections and infestations) | 12 (13) | 15 (16) | 5 (7)
Sinusitis (Infections and infestations) | 3 (5) | 5 (6) | 1 (1)
Tonsillitis (Infections and infestations) | 3 (3) | 6 (6) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 5 (7) | 19 (28) | 2 (6)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 6 (7) | 9 (12) | 1 (2)
Accidental Overdose (Injury, poisoning and procedural complications) | 2 (2) | 5 (5) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 1 (1)
Eyelid Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ligament Sprain (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 1 (1)
Wrist Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (4) | 8 (15) | 1 (1)
Tension Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 7 (10) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 2 (2)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT03560466/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT03560466/SAP_001.pdf